CLINICAL TRIAL: NCT04722276
Title: The Effect of Positive End-expiratory Pressure During Induction of General Anesthesia and Non-hypoxic Apnea Time in Infants: a Randomized Controlled Trials
Brief Title: Fraction of Oxygen on Induction of Anesthesia in Infants
Acronym: PEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-152-1184
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fraction of inspired oxygen 80% (Active Comparator)
  Interventions: Other: fraction of inspired oxygen 80%
- Fraction of inspired oxygen 80% with positive end expiratory pressure (Experimental)
  Interventions: Other: positive end expiratory pressure

INTERVENTIONS:
Other: positive end expiratory pressure — 7cmH2O of positive end expiratory pressure with fraction of inspired oxygen 80% applied during induction of anesthesia
  Arms: Fraction of inspired oxygen 80% with positive end expiratory pressure
Other: fraction of inspired oxygen 80% — fraction of inspired oxygen 80% applied during induction of anesthesia
  Arms: fraction of inspired oxygen 80%

SUMMARY:
Invesetigators evaluated the effect of positive end-expiratory pressure during anaesthesia induction on nonhypoxic apnoea time in infants. Invesetigators assigned infants to a 7 cmH2O positive end expiratory pressure (PEEP) with fraction of inspired oxygen 80% or 0 cmH2O PEEP with fraction of oxygen 80% group. Anaesthesia was induced with 0.02 mg kg atropine, 5 mg kg thiopental sodium and 3 to 5% sevoflurane, and neuromuscular blockade with 0.6 mg kg rocuronium. Thereafter, 80% oxygen was provided via face mask with volume-controlled ventilation of 6 ml kg tidal volume, and either 7 cmH2O or no positive end-expiratory pressure. After 3 min of ventilation, the infants' trachea was intubated but disconnected from the breathing circuit, and ventilation resumed when pulse oximetry reached 95%.

ELIGIBILITY:
Inclusion Criteria:

* We included paediatric patients aged 12 months or less about to receive general anaesthesia with endotracheal intubation.

Exclusion Criteria:

* Neonates, former preterm infants with gestational age less than 60 weeks at the day of surgery, with previous history of respiratory disease, those with anticipated difficult mask ventilation or intubation and those with upper respiratory infection within 3 weeks were excluded.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
apnea time | during face mask ventilation, maximum 3 minutes.
  The primary outcome was nonhypoxic apnoea time defined as the time from cessation of ventilation to a pulse oximeter reading of 95%

SECONDARY OUTCOMES:
atelectasis score (0~72) | during anesthesia induction, maximum 5 minutes.
  atelectasis score assessed by lung ultrasound (0-72)
Number of participants with gastric air insufflation | during anesthesia induction, maximum 5 minutes.
  presence of air in the gastric antrum

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea